CLINICAL TRIAL: NCT00631319
Title: A Phase III, Flexible Dose Titration Followed by a Randomized Double-Blind Study of Controlled Release OROS Hydromorphone HCL Compared to Placebo in Patients With OA Pain
Brief Title: A Double-blind Study of Controlled Release OROS Hydromorphone Compared to Placebo in Patients With Chronic Osteoarthritis (OA) Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NMT 1077-302
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Results first posted 2020-08-26 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-08

CONDITIONS: Chronic Pain
Keywords: OA; Chronic Pain; Osteoarthritis; OA Pain; Osteoarthritis Pain; Pain; Hip Pain; Knee Pain; Joint Pain
MeSH Terms: conditions — Chronic Pain; Osteoarthritis; Pain; Arthralgia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- OROS Hydromorphone (Experimental): OROS hydromorphone tablets administered orally once daily in total daily doses of 12, 16, 24, 32, 40, 48, or 64 mg
  Interventions: Drug: OROS hydromorphone
- Placebo (Placebo Comparator): Matching placebo tablets orally once daily (number and dosage of tablets to match the number and dosage of the stable dose of OROS hydromorphone obtained in the Conversion and Titration phase).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OROS hydromorphone — hydromorphone 12, 16, 24, 32, 40, 48, or 64 mg tablets
  Arms: OROS Hydromorphone
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
To evaluate the efficacy of OROS Hydromorphone in reducing moderate to severe chronic pain in patients with Osteoarthritis (OA) Pain

ELIGIBILITY:
Inclusion Criteria

* Primary clinic diagnosis of osteoarthritis pain of the hip or of the knee for at least 6 months
* Patients required daily opioid medication to treat their chronic osteoarthritis pain

Exclusion Criteria

* Joint replacement of the hip or of the knee that is the primary source of osteoarthritis Pain
* History drug or alcohol abuse
* Fibromyalgia
* Patients who have major depression or anxiety
* Women who are pregnant or breast feeding

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2008-02; Primary Completion 2009-04 (Actual); Study Completion 2009-06 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Matching placebo tablets orally once daily
Period: Conversion and Titration Phase
Arm/Group | OROS Hydromorphone | Placebo
Started | 343 | 0 (Per the study design, no patients received placebo during this phase.)
Completed | 200 | 0
Not Completed | 143 | 0
Period: Double-blind Phase
Arm/Group | OROS Hydromorphone | Placebo
Started (Patients who completed titration and conversion were allowed in the double-blind phase.) | 100 | 100
Completed | 60 | 65
Not Completed | 40 | 35

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OROS Hydromorphone | Placebo | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 83 | 77 | 160
  >=65 years | 17 | 23 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (9.78) | 55.4 (11.1) | 55.8 (10.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 53 | 107
  Male | 46 | 47 | 93
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 100 | 100 | 200

OUTCOME MEASURES:

1. Primary Outcome: Patient Diary-derived Numeric Rating Scale (NRS) Pain Intensity Change From Baseline to Week 12 or Final Visit of the Double-blind Phase
Description: Participants rate their pain intensity on a numeric rating scale (NRS), where 0=no pain and 10=worst possible pain, in a daily diary. At Week 12 (or final visit), all measurements during the preceding week are averaged, and the mean change from the mean score at baseline is calculated.
Time Frame: Baseline, Week 12
Population: Intent to treat population defined as all patients randomized to the Double-blind phase who received at least one dose of randomized study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- OROS Hydromorphone: OROS hydromorphone tablets administered orally once daily in total daily doses of 12, 16, 24, 32, 40, 48, or 64
Arm/Group | OROS Hydromorphone | Placebo
Number analyzed (Participants) | 100 | 100
units on a scale | 0.6 (2.02) | 0.6 (1.87)

2. Other Pre Specified Outcome: Patient Diary-derived Numeric Rating Scale (NRS) Pain Intensity and Change From Baseline by Visit in the Double-blind Phase
Time Frame: Baseline to Week 12
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score and Change From Baseline by Visit in the Double-blind Phase
Time Frame: Baseline to Week 12
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Stiffness Subscale Score and Change From Baseline by Visit in the Double-blind Phase
Time Frame: Baseline to Week 12
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscale Score and Change From Baseline by Visit in the Double-blind Phase
Time Frame: Baseline to Week 12
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Patient Global Assessment and Change From Baseline by Visit in the Double-blind Phase
Time Frame: Baseline to Week 12
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Time to Treatment Failure From Baseline
Time Frame: within 12 weeks from Baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Duration of the trial: 1 year, 4 months
Description: The safety population includes all patients who were enrolled and who took at least one dose of study drug (N=338). Adverse event displays include data from the safety population. The number of subjects who entered the Conversion and Titration phase was 343.
Groups:
- Conversion and Titration Phase; Double-blind Phase - Hydromorphone: OROS hydromorphone 12, 16, 24, 32, 40, 48 or 64 mg
- Double-blind Phase - Placebo: Matching placebo tablets orally once daily
Arm/Group | Conversion and Titration Phase | Double-blind Phase - Hydromorphone | Double-blind Phase - Placebo
Serious Adverse Events (participants affected / at risk) | 6/338 | 5/100 | 1/100
Other Adverse Events (participants affected / at risk) | 197/338 | 68/100 | 52/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Conversion and Titration Phase (N=338) | Double-blind Phase - Hydromorphone (N=100) | Double-blind Phase - Placebo (N=100)
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Gastroenteritis (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Drug toxicity (Injury, poisoning and procedural complications) | 1 | 0 | 0
Chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Completed suicide (Psychiatric disorders) | 1 | 0 | 0
Urethral caruncle (Renal and urinary disorders) | 1 | 0 | 0
Embolism (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Conversion and Titration Phase (N=338) | Double-blind Phase - Hydromorphone (N=100) | Double-blind Phase - Placebo (N=100)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 7 | 1
Constipation (Gastrointestinal disorders) | 59 | 20 | 4
Diarrhoea (Gastrointestinal disorders) | 0 | 6 | 7
Dry mouth (Gastrointestinal disorders) | 0 | 2 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 53 | 14 | 5
Toothache (Gastrointestinal disorders) | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 19 | 9 | 5
Drug withdrawal syndrome (General disorders) | 15 | 5 | 8
Fatigue (General disorders) | 11 | 2 | 1
Oedema peripheral (General disorders) | 10 | 4 | 1
Pyrexia (General disorders) | 0 | 2 | 3
Bronchitis (Infections and infestations) | 0 | 0 | 3
Gastroenteritis (Infections and infestations) | 0 | 4 | 0
Influenza (Infections and infestations) | 0 | 2 | 3
Nasopharyngitis (Infections and infestations) | 0 | 4 | 2
Sinusitis (Infections and infestations) | 9 | 3 | 2
Tooth abscess (Infections and infestations) | 0 | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 7 | 4 | 2
Urinary tract infection (Infections and infestations) | 0 | 3 | 3
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 2 | 0
Weight decreased (Investigations) | 0 | 3 | 2
Arthralgia (Metabolism and nutrition disorders) | 7 | 7 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 2 | 2
Joint stiffness (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Dizziness (Nervous system disorders) | 15 | 4 | 0
Headache (Nervous system disorders) | 22 | 5 | 7
Somnolence (Nervous system disorders) | 28 | 1 | 2
Tremor (Nervous system disorders) | 0 | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 8 | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No